CLINICAL TRIAL: NCT03458468
Title: A Randomised, Prospective Evaluation on the Effectiveness of Tranexamic Acid in Reducing Postoperative Swelling and Haematoma Formation After the Latarjet Procedure.
Brief Title: Tranexamic Acid for the Latarjet Procedure.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sports Surgery Clinic, Santry, Dublin (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SSC-Latarjet-001
Record Dates: First submitted 2018-02-19; First posted 2018-03-08 (Actual); Last update posted 2019-07-30 (Actual); Status verified 2019-07

CONDITIONS: Anterior Shoulder Instability
Keywords: tranexamic acid; anterior shoulder instability; latarjet; hematoma
MeSH Terms: conditions — Hematoma | interventions — Tranexamic Acid; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Double-blinded randomized
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Experimental): Tranexamic Acid 1g IV
  Interventions: Drug: Tranexamic Acid
- Group B (Placebo Comparator): Saline injection
  Interventions: Drug: Saline

INTERVENTIONS:
Drug: Tranexamic Acid — 1g Tranexamic acid prior to skin incision
  Arms: Group A
Drug: Saline — Equivalent volume of saline prior to skin incision
  Arms: Group B

SUMMARY:
The investigators propose a double-blinded randomized study evaluating the effectiveness of tranexamic acid in reducing postoperative swelling and haematoma formation after the Latarjet procedure.

The purpose of this study is to assess the efficacy of tranexamic acid (TXA), given via intra-articular injection at the time of surgery in patients undergoing the Latarjet procedure for shoulder instability.

ELIGIBILITY:
Inclusion Criteria:

• Anterior shoulder instability, warranting the Latarjet procedure

Exclusion Criteria:

* Patients with known risk factors for hyper-coagulable state
* Patients under 16
* Patients unable to give consent to partake in the trial

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2018-03-01 (Actual); Primary Completion 2019-03-01 (Actual); Study Completion 2019-03-01 (Actual)

PRIMARY OUTCOMES:
Hematoma Formation | Postoperative day-1
  Patients hematoma formation will be evaluated using the Pauzenberger criteria (Grade 1-4)
Visual Analogue Scale | Postoperative day-1
Total Drain output | Postoperative day-1
  The total drain output of blood post-operatively
Opioid consumption | Postoperative day-1

SECONDARY OUTCOMES:
Wound complications | Postoperative week-2
Total complications | Postoperative month-4
Haematoma Formation | Postoperative week-2

CONTACTS AND LOCATIONS:
Overall Officials: Hannan Mullett, FRCSI, Principal Investigator — Sports Surgery Clinic
Locations (1):
- Sports Surgery Clinic, Santry, Dublin, Ireland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Gillespie R, Shishani Y, Joseph S, Streit JJ, Gobezie R. Neer Award 2015: A randomized, prospective evaluation on the effectiveness of tranexamic acid in reducing blood loss after total shoulder arthroplasty. J Shoulder Elbow Surg. 2015 Nov;24(11):1679-84. doi: 10.1016/j.jse.2015.07.029. PMID 26480877
- [Background] Pauzenberger L, Domej MA, Heuberer PR, Hexel M, Grieb A, Laky B, Blasl J, Anderl W. The effect of intravenous tranexamic acid on blood loss and early post-operative pain in total shoulder arthroplasty. Bone Joint J. 2017 Aug;99-B(8):1073-1079. doi: 10.1302/0301-620X.99B8.BJJ-2016-1205.R1. PMID 28768785
- [Background] Vara AD, Koueiter DM, Pinkas DE, Gowda A, Wiater BP, Wiater JM. Intravenous tranexamic acid reduces total blood loss in reverse total shoulder arthroplasty: a prospective, double-blinded, randomized, controlled trial. J Shoulder Elbow Surg. 2017 Aug;26(8):1383-1389. doi: 10.1016/j.jse.2017.01.005. Epub 2017 Feb 3. PMID 28162887
- [Background] Kirsch JM, Bedi A, Horner N, Wiater JM, Pauzenberger L, Koueiter DM, Miller BS, Bhandari M, Khan M. Tranexamic Acid in Shoulder Arthroplasty: A Systematic Review and Meta-Analysis. JBJS Rev. 2017 Sep;5(9):e3. doi: 10.2106/JBJS.RVW.17.00021. PMID 28902659